CLINICAL TRIAL: NCT06388161
Title: Neural Autoantibody Prevalence in Patients With New-onset Focal Seizures of Unknown Etiology and a Predictive Scoring Scale
Brief Title: Neural Autoantibody Prevalence in New-onset Focal Seizures of Unknown Etiology
Status: Recruiting | Type: Observational
Sponsor: Shen Chun-Hong (Other)
Responsible Party: Sponsor-Investigator, Shen Chun-Hong, Associate Senior Doctor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Other Study IDs: Yan2022-0336
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy; Encephalitis Autoimmune
MeSH Terms: conditions — Epilepsy; Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum and cerebrospinal fluid samples will be stored to test antibodies, cytokines, and other relevant molecules. And patients have the right to destroy them at any time.
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Seizure is one of the most common symptoms in autoimmune encephalitis with neuronal surface-mediated antibodies. Interestingly, some patients may exhibit new-onset seizures as the initial manifestation without fulminant sign of encephalitis, particularly in the early stage.

It is essential to recognize these patients early and to perform antibody testing, as studies have reported early immunotherapy can improve their clinical outcomes. At the same time, it is important to limit the number of patients who require testing, for the sake of specificity and cost effectiveness. Thus, this prospective, multicenter study aims to identify neural antibodies in patients with focal seizures of unknown etiology, and to create a score to preselect patients requiring autoantibody testing.

DETAILED DESCRIPTION:
1. Focal epileptic seizure or epilepsy is defined according to seizure semiology, electroencephalography findings and/or other relevant information. If applicable, 24 hour video-electroencephalography is performed.
2. Clinical information is documented by specially-assigned persons, including patient demographics, age at onset, disease duration, seizure semiology, seizure frequency, clinical manifestations, underlying malignancy, hyponatremia, brain MRI, medications and other diseases.
3. The Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Hamilton Depression Scale (HAMA), Hamilton Anxiety Scale (HAMA) and the modified Rankin Scale (mRS) at baseline were assessed and recorded.
4. Previous scoring scales, such as antibody prevalence in epilepsy and encephalopathy (APE2) score, antibodies contributing to focal epilepsy signs symptoms (ACES) score and the "Obvious" Indications for Neural Antibody Testing in Epilepsy or Seizures (ONES) checklist are evaluated at baseline.
5. Commercial cell-based assay (CBA; EUROIMMUN, Lübeck, Germany) was used to detect serum anti-N-methyl-D-aspartate receptor (anti-NMDAR), anti-α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid receptor (anti-AMPAR), anti-γ-aminobutyric acid B receptor (anti-GABABR), anti-leucine-rich glioma-inactivated 1 (anti-LGI1), anti-contactin-associated protein-like 2 (anti-CASPR2), and anti-glutamic acid decarboxylase 65 (anti-GAD65), anti-metabotropic glutamate receptor 5 (mGluR5), anti-dipeptidyl peptidase-like protein 6 (DPPX), anti-myelin oligodendrocyte glycoprotein (MOG) and anti-immunoglobulin-like cell adhesion molecule 5 (IgLON5) antibodies. If serum neural autoantibodies are detected, cerebrospinal fluid should be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of new-onset focal epileptic seizure or epilepsy and present with their first seizure within the previous 12 months
* Patients are prospectively recruited from the routine practice of epileptologists in epilepsy centers and epilepsy clinics
* There is no obvious suspicion of autoimmune encephalitis
* Written informed consent and sera are obtained
* Cerebrospinal fluid test must be conducted, when patients have detectable serum autoantibodies

Exclusion Criteria:

* Patients have other etiology of seizures, such as structure, infection, genetics and metabolism.
* Written informed consent are not obtained
* Loss of follow-up

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have new-onset focal seizure with unknown etiology; and focal seizure is considered according to the seizure seiology, electroencephalography findings and/or other relevant information.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Detectable serum neural autoantibodies | at baseline
  such as NMDAR、AMPAR1、AMPAR2、LGI1、lg LON5、DPPX、GAD65、mGluR5、MOG
Neuronal surface antibodies-mediated autoimmune- encephalitis | at baseline
  diagnosed according to the 2016 diagnostic criteria

SECONDARY OUTCOMES:
The proportion of seizure freedom | through study completion, an average of 1 year
  We defined seizure freedom according to the International League Against Epilepsy (ILAE) definition
The proportion of drug-resistent epilepsy | through study completion, an average of 1 year
  We defined drug-resistent epilepsy according to the International League Against Epilepsy (ILAE) definition
Clinical severity and recovery | through study completion, an average of 1 year
  modified Rankin scale, ranging from 0-6, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chunhong Shen, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No